CLINICAL TRIAL: NCT00206882
Title: The Sun Protection Effect and Efficacy in Treatment of Sunburn Using Topical Corticosteroids.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Bispebjerg Hospital (Other)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: KF-01-272662
Record Dates: First submitted 2005-09-12; First posted 2005-09-21 (Estimated); Last update posted 2006-10-11 (Estimated); Status verified 2005-08

CONDITIONS: Sunburn
Keywords: sunburn; corticosteroids
MeSH Terms: conditions — Sunburn | interventions — Adrenal Cortex Hormones

INTERVENTIONS:
Drug: corticosteroids

SUMMARY:
The purpose of the study is to evaluate the sun protection effect and efficacy in treatment of sunburn using topical corticosteroids in a randomised controlled and investigator blinded trial.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older, healthy, fair skinned (skin type I-III)

Exclusion Criteria:

* Pregnant or lactating women.In treatment with corticosteroids.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20
Dates: Start 2005-09

CONTACTS AND LOCATIONS:
Overall Officials: Hans Christian Wulf, M.D., Dr.Sc., Study Director — Bispebjerg Hospital
Locations (1):
- Bispebjerg Hospital, Copenhagen, Copenhagen NV, Denmark

REFERENCES:
- [Derived] Faurschou A, Wulf HC. Topical corticosteroids in the treatment of acute sunburn: a randomized, double-blind clinical trial. Arch Dermatol. 2008 May;144(5):620-4. doi: 10.1001/archderm.144.5.620. PMID 18490588